CLINICAL TRIAL: NCT05704192
Title: Non-invasive CT-based Hepatic Venous Pressure Gradient Assessment for Predicting the Prognosis of Hepatocellular Carcinoma With Transarterial Chemoembolization (CHANCE-CHESS 2302): A Multicenter Retrospective Study
Brief Title: CT-based HVPG Assessment for Predicting the Prognosis of HCC With TACE (CHANCE-CHESS 2302)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, President, Zhongda Hospital
Other Study IDs: CHANCE-CHESS 2302
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma; Portal Hypertension
Keywords: hepatocellular carcinoma; transarterial chemoembolization; portal hypertension; non-invasive imaging assessment; deep learning
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinically significant portal hypertension (CSPH) group: A CT-based HVPG Score, whose computed formula was: 17.37-4.91*ln(Liver/Spleen volume ratio) +3.8[If presence of peri-hepatic ascites],was used to diagnose CSPH (HVPG>10mmHg) with a cut-off value 11.606.
  Interventions: Procedure: TACE ± Systemic therapy
- non-CSPH group: A CT-based HVPG Score, whose computed formula was: 17.37-4.91*ln(Liver/Spleen volume ratio) +3.8[If presence of peri-hepatic ascites],was used to diagnose CSPH (HVPG>10mmHg) with a cut-off value 11.606.
  Interventions: Procedure: TACE ± Systemic therapy

INTERVENTIONS:
Procedure: TACE ± Systemic therapy — TACE: conventional TACE (cTACE) or drug-eluting beads TACE (dTACE); Systemic therapy: programmed cell death protein-1 (PD-1)/programmed cell death ligand-1 (PD-L1) inhibitors, vascular endothelial growth factor -tyrosine kinase inhibitor (VEGF-TKI)/bevacizumab, PD-1/PD-L1 inhibitors+VEGF-TKI/bevacizumab, radiotherapy or chemotherapy.

SUMMARY:
This study aims to evaluate the impact of non-invasive CT-based Hepatic Venous Pressure Gradient (HVPG) assessment on prognosis of hepatocellular carcinoma (HCC) patients treated with transarterial chemoembolization (TACE).

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most common cancer worldwide and the second leading cause of cancer-related deaths globally. Transarterial chemoembolization (TACE) is recommended as standard therapy for intermediate-stage HCC according to the current guidelines and is also the most widely used in advanced HCC in real-world practice. Portal hypertension increases the risk of hepatic decompensation, which impairs survival in patients with HCC. Clinically significant portal hypertension is defined as >10 mmHg increase in the hepatic vein pressure gradient (HVPG), and the current gold standard for its assessment is direct measurement, through a transjugular approach. However, due to its invasive character and high effort, HVPG measurement is not a standard tool in the initial diagnostic evaluation of patients with HCC. This study aims to evaluate the impact of non-invasive CT-based Hepatic Venous Pressure Gradient (HVPG) assessment on prognosis of hepatocellular carcinoma (HCC) patients treated with transarterial chemoembolization (TACE).

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of HCC confirmed by radiology, histology, or cytology;
2. Received at least 1 TACE treatment；
3. Contrast-enhanced computed tomography (CECT) examination within 1 month before the first TACE treatment;

Exclusion Criteria:

1. Cholangiocarcinoma, fibrolamellar, sarcomatoid hepatocellular carcinoma, and mixed hepatocellular/cholangiocarcinoma subtypes(confirmed by histology, or pathology) are not eligible;
2. Eastern Cooperative Oncology Group - Performance Status (ECOG-PS) > 2;
3. History of liver or spleen resection;
4. Loss to follow-up;
5. CECT image data was incomplete, unclear, or artifact occurred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC treated with TACE ± Systemic Treatment from January 2010 to December 2021.
Sampling Method: Probability Sample
Enrollment: 373 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | up to approximately 2 years
  The OS is defined as the time from the initiation of any treatment to death due to any cause.

SECONDARY OUTCOMES:
Objective response rate(ORR) per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | up to approximately 2 years
  The ORR is defined as the proportion of patients with a documented complete response(CR) or partial response(PR) per mRECIST.
Progression free survival(PFS) per mRECIST | up to approximately 2 years
  The PFS is defined as the time from the initiation of any treatment to the first documented progressive disease (according to mRECIST) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Principal Investigator — Zhongda hospital, Southeast university, Nanjing, China; Xiaolong Qi, M.D., Principal Investigator — Zhongda Hospital, Medical School, Southeast University, Nanjing, China
Locations (2):
- China (2):
  - Gao-Jun Teng, Nanjing
  - Xiaolong Qi, Nanjing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller L, Hahn F, Mahringer-Kunz A, Stoehr F, Gairing SJ, Foerster F, Weinmann A, Galle PR, Mittler J, Pinto Dos Santos D, Pitton MB, Duber C, Fehrenbach U, Auer TA, Gebauer B, Kloeckner R. Prevalence and clinical significance of clinically evident portal hypertension in patients with hepatocellular carcinoma undergoing transarterial chemoembolization. United European Gastroenterol J. 2022 Feb;10(1):41-53. doi: 10.1002/ueg2.12188. Epub 2021 Dec 16. PMID 34918471
- [Background] Iranmanesh P, Vazquez O, Terraz S, Majno P, Spahr L, Poncet A, Morel P, Mentha G, Toso C. Accurate computed tomography-based portal pressure assessment in patients with hepatocellular carcinoma. J Hepatol. 2014 May;60(5):969-74. doi: 10.1016/j.jhep.2013.12.015. Epub 2013 Dec 19. PMID 24362073
- [Background] Yu Q, Huang Y, Li X, Pavlides M, Liu D, Luo H, Ding H, An W, Liu F, Zuo C, Lu C, Tang T, Wang Y, Huang S, Liu C, Zheng T, Kang N, Liu C, Wang J, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Fang Q, Fu CC, Zhang R, Wang C, Wei J, Tian J, Ormeci N, Ellik Z, Asiller OO, Ju S, Qi X. An imaging-based artificial intelligence model for non-invasive grading of hepatic venous pressure gradient in cirrhotic portal hypertension. Cell Rep Med. 2022 Mar 15;3(3):100563. doi: 10.1016/j.xcrm.2022.100563. eCollection 2022 Mar 15. PMID 35492878
- [Background] Faitot F, Allard MA, Pittau G, Ciacio O, Adam R, Castaing D, Cunha AS, Pelletier G, Cherqui D, Samuel D, Vibert E. Impact of clinically evident portal hypertension on the course of hepatocellular carcinoma in patients listed for liver transplantation. Hepatology. 2015 Jul;62(1):179-87. doi: 10.1002/hep.27864. Epub 2015 May 20. PMID 25914217